CLINICAL TRIAL: NCT03542396
Title: ImPuls - a Group Therapeutic Exercise Intervention for the Outpatient Psychotherapeutic Context
Brief Title: Evaluation of a Group Therapeutic Exercise Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ImPuls_2018
Record Dates: First submitted 2018-04-25; First posted 2018-05-31 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2019-12

CONDITIONS: Depression; Anxiety Disorders; Primary Insomnia; ADHD
Keywords: Behaviour change techniques; Aerobic exercise; Mental disorders
MeSH Terms: conditions — Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders; Attention Deficit Disorder with Hyperactivity; Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ImPuls (Experimental): Participants receive an supervised exercise intervention and behaviour change techniques for 4 weeks and, after that, they are encouraged to engage in physical activity for 8 weeks independently. During this 8-week individual phase, patients have weekly phone contacts with a psychotherapist
  Interventions: Behavioral: ImPuls
- Control (No Intervention): Participants do not receive any intervention. Participants receive treatment as usual, which means they are on a waiting list of an outpatient unit to receive individual psychotherapeutic treatment

INTERVENTIONS:
Behavioral: ImPuls — Participants receive an supervised exercise intervention and behaviour change techniques for 4 weeks and, after that, they are encouraged to engage in physical activity for 8 weeks independently. During this 8-week individual phase, patients have weekly phone contacts with a psychotherapist
  Arms: ImPuls

SUMMARY:
Moderate to vigorous physical activity can reduce symptoms of mental disorders like major depression, anxiety disorders, insomnia, and ADHD. However, in Germany there are no group therapeutical exercise programs for psychotherapy patients in an outpatient context. The current study aims to examine the effectiveness of a manualized exercise program, named ImPuls, which consists of a supervised and non-supervised endurance training in moderate to vigorous intensity and behaviour change techniques.

DETAILED DESCRIPTION:
The current study aims to examine the efficacy (i.e., symptom reduction, increase of heart rate variability, improvement of sleep quality, increase of intrinsic motivation to engage in physical activity, increase of the level of physical activity) of a three-months manualized group exercise program, named ImPuls. The program contains supervised and non-supervised endurance training combined with behaviour change techniques. The manual was designed for patients with major depression, anxiety disorders, insomnia, and ADHD who are waiting for psychotherapeutic treatment. It is assumed that the program will improve the psychopathological symptoms of the different mental disorders. Heart rate variability, level of exercise, sleep quality, motivation and symptoms are measured by objective measures (physiological measurements, accelerometers) and subjective measures (structured interviews and questionnaires). In a randomized controlled trial, ImPuls will be evaluated (n = 38 intervention group vs. n = 37 control group). For four weeks, small group sessions of three to four people take place three times a week, combining endurance exercise (i.e., running) and behaviour change techniques, supervised by two therapists. The training is based on the actual evidence for effective therapeutic effects on psychopathological symptoms, individually adapted to each patient's fitness level (60-80% of the maximal heart rate) and lasts 30 minutes. In the following eight weeks, participants are encouraged to engage in physical activity independently for two to three times a week. It is assumed that the program will reduce symptoms of the different mental disorders as well as increase the heart rate variability, improve sleep quality, intrinsic motivation to engage in physical activity, and the engagement in physical activity. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a primary DSM-5 diagnosis of depression (F32, F33, F34.1), anxiety disorder (F40- F44), ADHD (F90) or sleep disorders (F51)
* Participants must be aged between 18 and 65 years
* Have not changed their psychotropic drugs intake within the last two months
* Must be physically healthy on the basis of a medical examination
* Fluent in German
* Must be waiting for psychotherapy (waiting list)

Exclusion Criteria:

* Acute and remitted eating disorders (F50)
* Antisocial personality disorder (F60.2) and borderline personality disorder (F60.3)
* current alcohol or substance use disorder (dependence) (F10.2, F11.2, F12.2, F13.2, F14.2, F15.2, F16.2, F18.2, F19.2)
* current somatic symptom disorder with predominant pain (45.1)
* Lifetime Bipolar disorders (F31)
* Acute suicidality
* High fitness level (> 1x moderate physical activity (endurance training for at least 30 minutes / week)
* Having taken psychotropic drugs for less than two months
* Start of psychotherapy or any psychotropic drugs during the program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Symptom-Checklist-90®-Standard at Week 13 and one year after study completion | Baseline (week 0), posttreatment assessment (week 13), and follow-up assessment (one year after posttreatment assessment)
  The Symptom-Checklist-90®-Standard (SCL-90®-S, Franke, 2014) was used to identify participants' impairment of physical and mental symptoms. The SCL-90®-S is a self-report questionnaire which captures the subjectively perceived impairment of a person's physical and mental symptoms on various scales. For this study, the scales of Anxiety, Depression, Phobic anxiety, Uncertainty in social contact and compulsiveness were used. Symptoms are registered on a 5-point Likert-Scale ranging from 0 = "being no manifestation of symptoms" to 4 = "being a very strong manifestation of symptoms". Scores will be transformed into T-values with higher scores indicating increasing abnormality (A T-value ≥ 60 indicates clinical abnormality)

SECONDARY OUTCOMES:
Change from Baseline in Pittsburgh Sleep Quality Index at Week 13 and one year after study completion | Baseline (week 0), posttreatment assessment (week 13), and follow-up assessment (one year after posttreatment assessment)
  The Pittsburgh Sleep Quality Index (PSQI; Buysse et al., 1989) retrospectively measures sleep quality over the last four weeks. The components add up to a total score that can vary from 0 to 21, with a higher score indicating reduced sleep quality. A cut-off value of five allows a division into "good" and "bad" sleepers.
Change from Baseline in Sleep Questionnaire B - Revised version at Week 13 and one year after study completion | Baseline (week 0), posttreatment assessment (week 13), and follow-up assessment (one year after posttreatment assessment)
  With the self-report questionnaire Sleep Questionnaire B - Revised version (Schlaffragebogen B, SF-B/R; Görtelmeyer, 2011), the sleep behavior and sleep experience of the past two weeks can be described and assessed quantitatively and qualitatively. The questionnaire assesses the following 4 sleep indices: Difficulty to Fall Asleep and Difficulty to Sleep Through (1 = "no difficulties" to 4 = "severe and lasting difficulties"), Premature Awakening (1 = "no premature awakening" to 5 = "being severe and lasting premature awakening") and General Sleep Characterization (1 = "negative characterization" to 5 = "positive characterization"). The four scores (averages) range from 1 to 5 since the most scales follow this five-point format. Higher scores of the first three indices indicate more sleep difficulties whereas higher scores of the last index (General Sleep Characterization) indicate a better characterization.
Change from Baseline Score in Global Assessment of Functioning-Scale at Week 13 and one year after study completion | Baseline (week 0), posttreatment assessment (week 13), and follow-up assessment (one year after posttreatment assessment)
  The Global Assessment of Functioning-Scale (GAF-Skala; American Psychiatric Association, 2000) is a scale which is used to record the general functional level on axis V of the DSM-IV. On this scale, only the mental, social or professional functions are assessed. The Global Assessment of Functioning-Skala is used to track the clinical progress of patients. The rating is based on the therapist's evaluation. The patient can be asked optionally if the therapist is not sure about the patient's general function. Global functioning is registered on a scale of 1 to 100, with 1 being the lowest and 100 being the highest score of global functioning.
Change From Baseline in Perceived Stress Scale at Week 13 and one year after study completion | Baseline (week 0), posttreatment assessment (week 13), and follow-up assessment (one year after posttreatment assessment)
  The Perceived Stress Scale (PSS; Cohen, Kamarck, & Mermelstein, 1983) is the most widely used instrument to measure perceived stress. The self-assessment scale consists out of 10 items and measures the degree to which a situation is appraised as stressful on a 5-point Likert-Scale ranging from 0 = "never" to 4 = "very often". All items summed up build a total score indicating the level of perceived stress. Individual scores can range from 0 to 40 with higher scores indicating higher perceived stress.
Change from Baseline in Heart rate Variability at Week 13 and one year after study completion | Baseline (week 0), posttreatment assessment (week 13), and follow-up assessment (one year after posttreatment assessment)
  The heart rate variability (HRV) is an indicator for chronic stress and is measured by the ECG and activity sensor ekgMove (Movisens GmbH, Karlsruhe, Germany). HRV indices are the RMSSD (the square root of the squared mean of the sum of all differences of successive RR intervals) and the high frequency domain (HF; 0.15 - 0.4 Hz)
  measured by the ecg- and activity sensor ekgMove (Movisens GmbH, Karlsruhe, Deutschland). HRV indices are the RMSSD (the square root of the squared mean of the sum of all differences of successive RR intervals) and the high frequency domain (HF; 0.15 - 0.4 Hz)
Change From Baseline in German version of the 36-Item Short Form Health Survey at Week 13 and one year after study completion | Baseline (week 0), posttreatment assessment (week 13), and follow-up assessment (one year after posttreatment assessment)
  The 36-Item Short Form Health Survey (SF-36, Morfeld, Kirchberger, & Bullinger, 2011) is a self-report questionnaire which captures the quality of life of patients across eight dimensions of subjective health: Physical functioning, physical role function, physical pain, general health perception, vitality, social functioning, emotional role function and mental well-being. With a single item, the current state of health is also inquired in comparison to last year. For each variable item scores are coded, summed and transformed on to a scale from 0 (worst possible health state) to 100 (best possible health state).
Change From Baseline in the Physical Activity, Exercise, and Sport Questionnaire at Week 13 and one year after study completion | Baseline (week 0), posttreatment assessment (week 13), and follow-up assessment (one year after posttreatment assessment)
  The Physical Activity, Exercise, and Sport Questionnaire (Bewegungs- und Sportaktivitätfragebogen, BSA-F; Fuchs, Klaperski, Gerber, & Seelig, 2015) is a self-report questionnaire which measures physical activities in three areas: activity at work, leisure time activity and exercise activity. Participants are asked to specify whether they are currently performing one or more physical activities regularly and to indicate the frequency (per week) and the duration in minutes (per session) for each activity. Only activities that involve larger groups of skeletal muscles are considered to construct a Physical Activity Index (minutes of physical activity per week). The higher the Physical Activity Index the more the person engages in exercise activities.
Physical activity (objective) | week 9
  Differences of the physical activity level (moderate to vigorous intensity) using the accelerometer Move II ((Movisens GmbH, Karlsruhe, Germany).
Change From Baseline in Self Concordance of Sport- and Exercise-related Goals Scale at Week 5 and 13 and one year after study completion | Baseline (week 0), posttreatment assessment (week 13), and follow-up assessment (one year after posttreatment assessment)
  The Self Concordance of Sport- and Exercise-related Goals Scale (SKK-Scale, Seelig & Fuchs, 2006) is a self-report questionnaire which measures how strongly the athletic goal intention matches the person's personal interests and values. Four subscales with three items each indicate the intrinsic, identified, introjected and extrinsic motivation of being physically active. Response format is a 4-point-Likert-scale ranging from 1 = "not true" to 4 = "true". A general index for self-concordance of sport- and exercise-related goals (SKK index) will be formed by summing up the identified and intrinsic means scores and subtracting the introjected and extrinsic mean scores. The lowest possible index value is -10 and the highest is +10. A high positive value indicates a strong self-concordance.
Change From Baseline in self-efficacy at Week 5 and 13 and one year after study completion | Baseline (week 0), posttreatment assessment (week 13), and follow-up assessment (one year after posttreatment assessment)
  Three different scopes of exercise-related self-efficacy are assessed (vgl. Göhner, Seelig, & Fuchs, 2009). Each scope is measured by one item on a 6-point Likert-scale ranging from 0 = "I don't feel capable at all" to 5 = "I feel 100 per cent capable". The scores of each item will be combined into one mean value with higher scores indicating a stronger self-efficacy.
Change From Baseline in strength of goal intention at Week 5 and 13 and one year after study completion | Baseline (week 0), posttreatment assessment (week 13), and follow-up assessment (one year after posttreatment assessment)
  Strength of goal intention is assessed with one item (vgl. Göhner et al., 2009). Response format is a 6-point Likert-scale ranging from 0 = "I don't have this intention at all" to 5 = "I do have a strong intention". A higher score indicates a stronger goal intention.
Change From Baseline in implementation intentions at Week 5 and 13 and one year after study completion | Baseline (week 0), posttreatment assessment (week 13), and follow-up assessment (one year after posttreatment assessment)
  The self-report scale implementation intentions (vgl. Göhner et al., 2009) measures whether the person know which physical activity they plan to perform in the following time. A second activity can be named. If the answer is "yes", the person is asked to note the named activity or activities. Subsequently, participants are asked if they would already know the location and time they would perform it as well as how they would get there, how often and with whom they would perform this activity. Positive answers will be summed up to build a score for implementation intentions (including naming the activity and planning details). A higher score indicates stronger implementation intentions. The score can range from 0 to 12.
Change From Baseline in Volitional Intention Shielding at Week 5 and 13 and one year after study completion | Baseline (week 0), posttreatment assessment (week 13), and follow-up assessment (one year after posttreatment assessment)
  The index Volitional Intention Shielding (VIS-index, vgl. Göhner et al., 2009) consists of the subscales "Perceived Barriers" and "Counter Strategies". The subscale Perceived Barriers measures how strongly barriers keep the person from exercising. On a list with 19 possible barriers, the participant can indicate how strongly these barriers (on a 4-point Likert-scale ranging from 1 = "not at all" to 4 = "very much") keep him from exercising. The mean of the 19 scores build the subscale Perceived Barriers. The subscale Counter Strategies indicates possible ways to overcome those barriers. A list presents 15 possible counter strategies. Response format is dichotomous with 1 = "Yes, I use this strategy" and 0 = "No, I don't use this strategy". The subscale Counter Strategies is the mean of the 15 scores. The quotient of the two subscales builds the VIS-index (range 0-1). The higher the VIS-index, the more successful is the intention shielding.
Change From Baseline in Physical Activity-related Health Competence Questionnaire at Week 13 and one year after study completion | Baseline (week 0), posttreatment assessment (week 13), and follow-up assessment (one year after posttreatment assessment)
  The Physical Activity-related Health Competence Questionnaire (Sudeck & Pfeifer, 2016) is a self-report questionnaire which certain aspects of physical activity-related health competence on a Likert scale from 1 = "strongly disagree" to 4 = "strongly agree". Sub-competencies are 1) movement Competence (6 items), 2) Control Competence (3 items), and 3) Physical-activity-specific self-regulation competence (4 items). All items will be summed, and the total score indicates the level of physical activity-related health competence. Individual scores can range from 13 to 52 with higher scores indicating higher physical activity-related health competence.
Change from Baseline in the The Homburg's ADHS Scales for adults at Week 13 | Baseline (week 0) and posttreatment assessment (week 13)
  The Homburg's ADHS Scales for adults (Homburger ADHS-Skalen für Erwachsene, HASE; Rösler, Retz-Junginger, Retz, & Stieglitz, 2007) serves for the diagnosis of ADHD in adulthood.The instrument consists of four separate procedures. For the current study, two of them were used: (1) The Wender Utah Rating Scale - German version (WURS-K) is used for retrospective diagnosis of childhood ADHD symptoms.
  (2) The ADHD self-assessment scale (ADHD-SB) includes the 18 diagnostic criteria of DSM-IV and of the ICD-10 research version. The individual characteristics can be scaled from 0 to 3 with higher scores indicating a higher symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Wolf, Dr., Principal Investigator — University Hospital Tuebingen
Locations (1):
- University of Tubingen, Faculty of Science, Clinical Psychology and Psychotherapy, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Zeibig JM, Seiffer B, Sudeck G, Rosel I, Hautzinger M, Wolf S. Transdiagnostic efficacy of a group exercise intervention for outpatients with heterogenous psychiatric disorders: a randomized controlled trial. BMC Psychiatry. 2021 Jun 22;21(1):313. doi: 10.1186/s12888-021-03307-x. PMID 34158000